CLINICAL TRIAL: NCT01163201
Title: Optimization of the T Regulatory Cell and T Effector Cell Doses in Recipients of Double UCB Transplantation for Treatment of Hematological Malignancies
Brief Title: T-Regulatory Cell and CD3 Depleted Double Umbilical Cord Blood Transplantation in Hematologic Malignancies
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Replaced by a new study
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009LS018; MT2009-03 (Other: Blood and Marrow Transplantation Program); 0910M73595 (Other: IRB, University of Minnesota)
Record Dates: First submitted 2010-05-26; First posted 2010-07-15 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Hematologic Malignancy; Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Myelogenous Leukemia in Blast Crisis; Anemia, Refractory, With Excess of Blasts; Chronic Myeloproliferative Disease; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Marginal Zone B-cell Lymphoma; Follicular Lymphoma; Lymphoplasmacytic Lymphoma; Mantle-Cell Lymphoma; Prolymphocytic Lymphoma; Large Cell Non-Hodgkin's Lymphoma; Lymphoblastic Lymphoma; Burkitt's Lymphoma; High Grade Non-Hodgkin's Lymphoma
MeSH Terms: conditions — Hematologic Neoplasms; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Anemia, Refractory, with Excess of Blasts; Myeloproliferative Disorders; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Burkitt Lymphoma | interventions — fludarabine; fludarabine phosphate; Cyclophosphamide; Whole-Body Irradiation; Cord Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treg Plus CD3+Teff Treatment (Experimental): Includes dose adjustment of T regulatory (Treg) and CD3+ T effector (CD3+ Teff) cells in recipients of double UCB transplantation
  Interventions: Biological: Treg cells; Biological: CD3+ Teff cells; Drug: Fludarabine; Drug: Cyclophosphamide; Radiation: Total body irradiation; Biological: Umbilical cord blood transplantation

INTERVENTIONS:
Biological: Treg cells — Given by infusion on Day 0 after transplantation - Five doses of Treg (3 x 10^6/kg, 10 x 10^6/kg, 30 x 10^6/kg, 100 x 10^6/kg and 300 x 10^6/kg)
Biological: CD3+ Teff cells — Given by infusion on Day 0 after transplantation - 5 doses of CD3+ Teff cells (3 x 10^6 cells/kg, 6 x 10^6 cells/kg, 9 x 10^6 cells/kg, 12 x 10^6 cells/kg, and 15 x 10^6 cells/kg with the latter dose representing the median number of CD3+ cells in two UCB unit grafts
Drug: Fludarabine — Given intravenously on Days -8 through -6, 25 mg/m^2 over 1 hour
  Other Names: Fludara
Drug: Cyclophosphamide — Given intravenously on Day -7 and -6, 60 mg/kg
  Other Names: Cytoxan
Radiation: Total body irradiation — Given on Days -4 through -2, 165 cGY twice a day.
Biological: Umbilical cord blood transplantation — Infusion given on day 0
  Other Names: UCBT

SUMMARY:
This is a unique dose-escalation trial that will titrate doses of umbilical cord blood (UCB) Treg and CD3+ Teff cells with the goal of infusing as many CD3+ Teff cells as possible without conferring grade II-IV acute graft-versus-host disease (GVHD).

In this study, the investigators propose to add UCB Treg and UCB CD3+ Teff cells to the two TCD UCB donor units with the goal of transplanting as many CD3+ Teff cells as possible without reintroducing risk of acute GVHD. The investigators hypothesize that Treg will permit the reintroduction of CD3+ Teff cells that will provide a bridge while awaiting HSC T cell recovery long term. The co-infusion of Treg will prevent GVHD without the need for prolonged pharmacologic immunosuppression.

DETAILED DESCRIPTION:
Based on prior studies, the first patient will start at lowest dose combination (3 x 10^6/kg of Treg and 3 x 10^6/kg of CD3+ Teff cells).

One patient will be entered at each level with a minimum of 35 days to observe the patient prior to moving to the next dose level. (1) If GVHD does not occur, a "successful step", then the CD3+ Teff cell dose will increase to the next higher level for the next patient; (2) If GVHD occurs, a "failed step", then Treg dose will increase to the next higher level for the next patient. It would take a minimum of 5 (if no GVHD) and maximum of 9 patients (if GVHD is observed at each level) to complete all Treg:CD3+ Teff cell combinations.

An additional 10 patients will be enrolled to verify that this reflects the optimal combination and evaluate its safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Only patients requiring a double umbilical cord blood (UCB) transplant are to be considered for this study.

UCB Requirements

* Three UCB units are required - one for Treg production and two for UCB transplant. The unrelated UCB donors must be 4-6/6 HLA-A, B, DRB1 matched with the recipient (HLA matching using molecular techniques: A and B to antigen level resolution and DR to allele level resolution). Suitable UCB units will be selected according to the University Of Minnesota UCB Graft Selection Algorithm.
* Suitable UCB units must be ABO matched.

Disease Criteria:

* Patients aged 18 to 55 years
* Acute Myeloid Leukemia: with morphologically persistent disease in a representative bone marrow aspirate sample with ≤ 10% blasts after at least 1 cycles of chemotherapy (if patient refuses or is disqualified from alternative protocols), or in 3rd or higher complete remission (CR).
* Acute Lymphocytic Leukemia: with morphologically persistent disease in a representative bone marrow aspirate sample with ≤ 10% blasts after at least 1 cycles of chemotherapy, or in 3rd or higher CR
* Chronic Myelogenous Leukemia in Blast Crisis: with ≤10% residual blasts in the bone marrow aspirate after at least 1 cycle of induction chemotherapy in combination with a tyrosine kinase inhibitor (TKI)
* Refractory Anemia with Excess Blasts: (≤ 10%) in representative bone marrow aspirate sample of blasts after 1 cycle of induction chemotherapy. If treated with hypomethylating agents, patients are eligible if blast count is ≤ 10% after 4 cycles or evidence of stable or progressive disease after at least 2 cycles.
* Chronic Myeloproliferative Disease
* Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma, Marginal Zone B-Cell Lymphoma or Follicular Lymphoma: disease must be refractory after at least two chemotherapy regimens or is chemotherapy sensitive but has residual nodal disease of ≥ 5 cm
* Lymphoplasmacytic Lymphoma, Mantle-Cell Lymphoma, Prolymphocytic Leukemia: disease must be refractory after at least two chemotherapy regimens or is chemotherapy sensitive but has residual nodal disease of ≥ 5 cm
* Large Cell Non-Hodgkin's Lymphoma: disease must be refractory after at least two chemotherapy regimens or is chemotherapy sensitive but has residual nodal disease of ≥ 5 cm
* Lymphoblastic Lymphoma, Burkitt's Lymphoma, and other High-Grade NHL: disease must be refractory after at least two chemotherapy regimens or is chemotherapy sensitive but has residual nodal disease of ≥ 5 cm
* Performance Status, Age, and Organ Function
* Adequate performance status defined as a Karnofsky score ≥ 80%
* Adequate organ function defined as:

  * Renal: creatinine < 2.0 mg/dL,
  * Hepatic: bilirubin, AST/ALT, ALP < 5 x upper limit of normal,
  * Pulmonary function: DLCOcorr > 50% normal,
  * Cardiac: left ventricular ejection fraction > 45%
* Voluntary written informed consent signed before performance of any study-related procedure not part of normal medical care

Exclusion Criteria:

* Available medically suitable HLA-identical related donor
* Active infection at time of transplantation (including active infection with Aspergillus or other mold within 30 days)
* History of HIV infection
* Pregnant or breast feeding. The agents used in this study may be teratogenic to a fetus and there is no information on the excretion of agents into breast milk. Females of childbearing potential must have a blood test or urine study within 14 days prior to registration to rule out pregnancy
* Prior myeloablative transplant within the last 6 months
* Extensive prior therapy including > 12 months alkylator therapy or > 6 months alkylator therapy with extensive radiation
* Patients who have received Y-90 ibritumomab (Zevalin) or I-131 tositumomab (Bexxar) as part of their salvage therapy (not eligible for myeloablative umbilical cord blood transplant)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
Optimal Cell Dose Mixture | Day 0
  Determine the optimal cell dose mixture of UCB T regulatory and CD3+ T effector cells without the development of grade II-IV acute GVHD

SECONDARY OUTCOMES:
Determine incidence of infusional toxicity | 48 hours
  reaction that occurs with 48 hours of product infusion
Incidence of neutrophil recovery | Day 42
  Determine the incidence of neutrophil recovery (absolute neutrophil count ≥ 500/uL) at day 42
Incidence of double and single chimerism | Day +21, Day +180, 1 Year
  Determine incidence of double and single unit chimerism at various time points
Incidence of Viral and Fungal Infections | 1 Year
  Determine incidence of viral and fungal infections at 1 year
1 Year Survival | 1 Year
  Estimate the probability of survival at 1 year
Incidence of Grade III-IV Acute Graft-Versus-Host Disease | Day 100
  Determine the incidence of grade III-IV acute GVHD at day 100
Incidence of Treatment Related Death | 6 Months
  Determine the incidence of treatment related mortality (TRM) at 6 months
Incidence of Platelet Recovery | 1 Year
  Determine the incidence of platelet recovery (platelet count ≥ 50,000/uL) at 1 year
Incidence of Chronic Graft-Versus-Host Disease | 1 Year
  Determine the incidence of chronic GVHD at 1 year
Incidence of Relapse | 1 Year
  Determine the incidence of relapse at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States